CLINICAL TRIAL: NCT06261268
Title: Strip Graft With Xenogeneic Matrix Versus Free Gingival Graft for the Augmentation of Peri-implant Keratinized Mucosa: A Randomized Clinical Trial With Vascular Analysis
Brief Title: Strip Graft w/ Xenogeneic Matrix vs Free Gingival Graft for the Augmentation of Peri-implant Keratinized Mucosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Strip vs FGG
Record Dates: First submitted 2024-01-16; First posted 2024-02-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantational Loss; Surgical Wound; Healing Surgical Wounds; Thin-gingiva
Keywords: Strip graft; Free gingival graft; Peri-implant keratinized mucosa; Soft tissue augmentation; Early wound healing; Postoperative blood supply
MeSH Terms: conditions — Surgical Wound | interventions — Mucograft

STUDY DESIGN:
Intervention Model Description: A randomized controlled equivalence clinical trial will be performed, with two parallel groups, a 1:1 allocation ratio, and a 12-month follow-up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Strip graft with Mucograft (Experimental): An apically repositioned flap is prepared then, a free epithelialized gingival strip graft is harvested from the molar area of the palate and sutured to the apical part of the recipient area. A xenogeneic collagen matrix (Mucograft®. Geistlich Pharma AG, Wolhusen, Switzerland) covers the remaining uncovered part of the periosteal bed.
  Interventions: Procedure: Strip graft with Mucograft
- Free gingival graft (Active Comparator): Apically repositioned flap is prepared. An epithelialized free gingival graft is harvested from the molar area of the palate, and sutured to the recipient area
  Interventions: Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Strip graft with Mucograft — An apically repositioned flap is made in the vestibular region. The flap is then elevated with a split-thickness preparation, and the mucogingival junction will be repositioned apically and fixed with periosteal-anchored sutures. Then, a free epithelialized gingival strip graft will be harvested from the molar area of the palate. The "Strip" graft is sutured to the apical end of the recipient bed. The remaining uncovered part of the periosteal bed will be covered with a xenogeneic collagen matrix (Mucograft®. Geistlich Pharma AG, Wolhusen, Switzerland) fixed with simple interrupted and crossed sutures. The edges of the palatal wound (donor area) will be approximated with crossed sutures.
  Arms: Strip graft with Mucograft
Procedure: Free gingival graft — The preparation of the apically repositioned flap and the recipient bed with its apico-coronal design and dimension is performed as in the test group. Subsequently, an epithelialized free gingival graft with the size of the entire recipient area with a thickness of 2 mm will be harvested from the molar area of the palate. The graft is sutured to the recipient periosteal bed using simple interrupted and crossed sutures. In the donor area, a collagen sponge is sutured to the wound by means of crossed sutures.
  Arms: Free gingival graft

SUMMARY:
The primary objective of this study is to compare changes in peri-implant keratinized mucosa (PIKM) following the application of apically repositioned flap (ARF) using a combination of a Strip graft and a Xenogeneic matrix, or with a free gingival graft (FGG), in implants in the second stage with <2 mm of PIKM.

Additionally, as a secondary objective, the investigators compare postoperative blood supply in both recipient and donor sites based on the type of graft obtained. Meanwhile, the investigators evaluate differences between the two groups concerning microcirculation values (perfusion units, PU), soft tissue thickness (STT), volume change, vestibular depth, as well as clinical, aesthetic, and patient-reported outcome measures (PROMS).

DETAILED DESCRIPTION:
1. BACKGROUND The importance of keratinized tissue around teeth and dental implants is a frequently investigated topic in the literature. The need for an adequate amount of peri-implant keratinized mucosa (PIKM), which is defined as a minimum width of 2 mm is demonstrated according to a recently published systematic review and consensus report.

   The standard of care in the PIKM augmentation is the apically repositioned flap (ARF) combined with a free gingival graft (FGG), as it represents a predictable and documented strategy to gain KT width. However, such technique implies the harvest of abundant autogenous grafts, and is frequently associated to sub-optimal aesthetic results due to the poor color mimicry of the grafted tissue.

   In light of such limitations, some alternatives based on the use of soft tissue substitutes have been proposed, with the aim of reducing surgical invasiveness through the avoidance of large autogenous grafts and improving aesthetic outcomes.

   Among those, the sole use of as xenogeneic collagen matrices (XCM) has been associated with promising clinical outcomes albeit with lesser KT width gains as compared to autogenous FGGs.

   Recently, a novel approach called the Strip Technique (ST) has been introduced, where the exposed periosteal bed of a ARF is covered with the combination of a xenogeneic collagen matrix and a 2-3 mm wide strip of autogenous free gingival graft, sutured at the apical border of the matrix. The rationale for this "combined grafting technique" stands on reducing surgical invasiveness and improving color mimicry through the use of a XCM, while providing a source of autogenous keratinizing cells in the apical border of the grafted area to promote better PIKM gains. Albeit this new approach seems promising, there is limited evidence regarding its clinical efficacy and there is a lack of knowledge regarding how the adoption of such combined approach affects the re-perfusion of the grafted tissue and the overall microvascular healing of the surgical site.

   Furthermore, the pattern of the revascularization of both the autologous grafts and the XCM requires further understanding. Most of our recent knowledge comes from classical animal studies that evaluated the microvascularization of FGG when placed over periosteum with microscopy. The postoperative blood supply of these free grafts is of key importance to their survival.

   Recently a new non-invasive technique has been introduced in the field of medicine and dentistry the Laser Speckle Contrast Imaging (LSCI) system, that provides further understanding on the dynamics of postoperative blood supply of the applied grafts and elucidate regarding the healing pattern of the strip combination technique.
2. JUSTIFICATION There is a lack of knowledge regarding the clinical performance, the healing pattern and the dynamics of revascularization when performing apically repositioned flaps combined with either the autogenous strip-XCM technique or autogenous FGGs.

Results from this study could assess whether the strip-XCM technique represents a reliable, less invasive, and simplified alternative to autogenous FGGs for the increase of PIKM.

Moreover, it could provide additional knowledge regarding the healing and revascularization pattern of both strip-XCM and FGGs around dental implants, assessed through an innovative technology as Laser Speckle Perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Short-span dental implants in the mandible at second stage with inadequate PIKM (<2 mm) with at least one adjacent tooth mesially
* Periodontally healthy patients with a pristine or reduced periodontium
* Plaque index (FMPS) less than 20%.

Exclusion Criteria:

* Compromised general health status that contraindicates study procedures (≥ASA III);
* Drug or alcohol abuse;
* Smoking of > 10 cigarettes per day;
* Chronic use of corticosteroids, NSAIDs or immunomodulators (any type or dose);
* Pregnant or lactating women;
* History of previous mucogingival surgeries in the area of interest

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in peri-implant keratinized mucosa width (mm) | Baseline, 1, 3, 6 and 12 months
  the apico-coronal linear dimension of the buccal peri-implant keratinized mucosa (PIKM) will be measured with a UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA) as the linear dimension of the buccal vestibule, from the buccal peri-implant mucosa margin to the mucogingival junction at the mid-buccal aspect of the treated implant and adjacent mesial tooth.

SECONDARY OUTCOMES:
Vascularization (in Laser Speckle perfusion units [LSPU]) | pre-surgically, post-surgically at 4, 7, 10, 14 and 30 days, and at 3-6 and 12 months
  Vascularization will be measured using Laser Speckle Contrast Imaging (LSCI) (PeriCam PSI System; Perimed AB, Sweden). This novel technology represents a validated, non-invasive, real time, chair side mean to provide contrast based bi-dimensional representations of the superficial vascular network of a given tissue surface.
Changes in soft tissue thickness (STT) (mm) | Baseline, post-op, 1, 3, 6 and 12 months
  STT will be measured by ultrasonography with a dental Pirop® ultrasound device (Echoson Company, Poland). The equipment is validated in experimental and clinical studies. Patients will undergo a clinical and ultrasound examination before gingival augmentation, as well as right after the surgery, at 1, 3, 6 and 12 months after, in order to evaluate STT at two different apico-coronal location. It will be measured at the mid-buccal aspect of the implant. Point 1 will be located 2 mm from the periimplant mucosal margin and point 2 will be considered at the mucogingival junction (MGJ).
Vestibule depth (VD) (mm) | Pre-surgically, and at 30 days, 3-6 and 12 months
  VD will be measured with a UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA) as the linear dimension of the buccal vestibule. At the mid-buccal aspect of the treated implant from the peri-implant soft tissue margin to the greatest concavity of the vestibule crease, retracting the lips with a spandex retractor for intraoral photography
Probing pocket depth (PPD) (mm) | pre-surgically, at 3, 6 and 12 months after surgery
  Probing depth will be measured from the peri-implant mucosal margin to the bottom of the sulcus, at 6 locations per implant, using a UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA), approximating to the nearest 0.5 mm.
Dehiscence (mm) | post-surgically, at 3, 6 and 12 months after surgery
  Recession will be measured from the peri-implant mucosal margin to the top of the healing abutment, at 6 locations per implant, using a UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA), approximating to the nearest 0.5 mm.
Full-mouth plaque score (FMPS) | Baseline, 1 month, 3 months, 6 and 12 months
  Full-mouth plaque score (FMPS) will be measured using a calibrated UNC15 periodontal probe (UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA). Score will be expressed in percentage (%), it will be calculated by the number of sites where plaque is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the bleeding index as a percentage. 6 sites per tooth is recorded.
Volumetric changes | Baseline, 14 days, 1 month, 3, 6 and 12 months
  Changes in the peri-implant tissue volume distribution will be analyzed by digital volumetric analysis (DVA), comparing preoperative data with measurements collected at different time points. At each time point, the treated area will be optically scanned with a 3D scanner (Medit i500, Medit Corp., Seoul, South Korea) and standard tessellation language (STL) will be analyzed with a dedicated software (Smop® Swissmeda Software, Swissmeda AG, Zurich, Switzerland), to superimpose the digital models acquired at the different timepoints. For each overlay, a sagittal section perpendicular to the implant axis in its central part (largest diameter) will be selected. A line coincident with the longitudinal axis of the implant will then be drawn on the cross-sectional images of such section, and an image capture (ImageJ, National Institutes of Health, Maryland, USA) will be exported for horizontal measurements.
Patient reported outcome measures (PROMS) | immediately after the surgery, 12 hours after the surgery, 1 day, 2, 3, 4, 5, 6, 7 days and 2 weeks after the surgery
  Patients' pain and discomfort with respect to the procedure will be assessed on a visual analogue scale (VAS) (0-10 cm, where 0 is the worst and 10 is the best). In addition, patients will be asked to report the amount of paracetamol they have consumed for pain control each day during the first postoperative week. Patients will be asked to fill out an additional questionnaire at 6 months and 1 year about their perception of the treatment. Aspects will be as follows: comfort of the treated area (during mastication and brushing) and aesthetic.
Esthetic analysis | 30-day, 3-, 6- and 12-month
  An examiner blinded to the patient allocation will assess the 30-day, 3-, 6- and 12-month photographs to score the aesthetic outcome of the intervention in Visual Analogue Scale (VAS) (0-10cm, where 0 is the worst and 10 is the best). The following aspects will be evaluated: color matching, tissue blending and the satisfaction of the patient.
Intra-surgical parameters | During surgery
  Both the harvested grafts, the applied xenogeneic matrix' dimension and the prepared recipient site will be measured and documented during the surgery. The measurements will be done using a UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA), to the nearest 0.5 mm.
Intra-surgical time | During the surgery
  Surgical time will be recorded.
Demographic data | Baseline
  affiliation data (age and sex) is recorded. For age the birthdate is recorded.
Anamnesis data | Baseline, through study completion, an average of 1 year
  previous medical history (systemic diseases, medication, allergies)
Smoking habit | Baseline, through study completion, an average of 1 year
  Smoking habit is recorded in number of cigarettes per day.
Full-mouth bleeding score (FMBS) (%) | Baseline, 1 month, 3 months, 6 and 12 months
  Full-mouth bleeding score (FMBS) will be measured using a calibrated UNC15 periodontal probe (UNC15 periodontal probe (Hu-Friedy manufacturing, Co., LLC, Chicago, USA). Score will be expressed in percentage (%), it will be calculated by the number of sites where bleeding is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the bleeding index as a percentage. 6 sites per tooth is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Study Director — Universidad Complutense de Madrid
Locations (1):
- Complutense University, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramanauskaite A, Schwarz F, Sader R. Influence of width of keratinized tissue on the prevalence of peri-implant diseases: A systematic review and meta-analysis. Clin Oral Implants Res. 2022 Jun;33 Suppl 23:8-31. doi: 10.1111/clr.13766. PMID 35763022
- [Background] Sanz M, Schwarz F, Herrera D, McClain P, Figuero E, Molina A, Monje A, Montero E, Pascual A, Ramanauskaite A, Renouard F, Sader R, Schiegnitz E, Urban I, Heitz-Mayfield L. Importance of keratinized mucosa around dental implants: Consensus report of group 1 of the DGI/SEPA/Osteology Workshop. Clin Oral Implants Res. 2022 Jun;33 Suppl 23:47-55. doi: 10.1111/clr.13956. PMID 35763021
- [Background] Montero E, Molina A, Matesanz P, Monje A, Sanz-Sanchez I, Herrera D. Efficacy of soft tissue substitutes, in comparison with autogenous grafts, in surgical procedures aiming to increase the peri-implant keratinized mucosa: A systematic review. Clin Oral Implants Res. 2022 Jun;33 Suppl 23:32-46. doi: 10.1111/clr.13751. PMID 35763018
- [Background] Solonko M, Regidor E, Ortiz-Vigon A, Montero E, Vilchez B, Sanz M. Efficacy of keratinized mucosal augmentation with a collagen matrix concomitant to the surgical treatment of peri-implantitis: A dual-center randomized clinical trial. Clin Oral Implants Res. 2022 Jan;33(1):105-119. doi: 10.1111/clr.13870. Epub 2021 Oct 21. PMID 34651349
- [Background] Urban IA, Lozada JL, Nagy K, Sanz M. Treatment of severe mucogingival defects with a combination of strip gingival grafts and a xenogeneic collagen matrix: a prospective case series study. Int J Periodontics Restorative Dent. 2015 May-Jun;35(3):345-53. doi: 10.11607/prd.2287. PMID 25909521
- [Background] Molnar E, Molnar B, Lohinai Z, Toth Z, Benyo Z, Hricisak L, Windisch P, Vag J. Evaluation of Laser Speckle Contrast Imaging for the Assessment of Oral Mucosal Blood Flow following Periodontal Plastic Surgery: An Exploratory Study. Biomed Res Int. 2017;2017:4042902. doi: 10.1155/2017/4042902. Epub 2017 Jan 23. PMID 28232940
- See also: Institutional homepage — https://www.ucm.es/directorio/?eid=3214